CLINICAL TRIAL: NCT07101419
Title: Longer Pressure Rise Time During Mechanical Ventilation of Extremely Preterm Infants: A Randomised Crossover Trial
Brief Title: Speed of Lung Inflation During Ventilation of Extremely Preterm Infants
Acronym: FLOW-VENT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: Mercy Hospital for Women, Australia (Other); Royal Women's Hospital, Melbourne, Australia (Unknown); Western Health, Australia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 117784
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome in Premature Infant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn

STUDY DESIGN:
Intervention Model Description: Extremely preterm infants on synchronised, patient-triggered, volume targeted conventional mechanical ventilation are managed with each pressure rise time (PRT) setting for 4 hours (treatment period 1), prior to crossing over to the other PRT setting for a further 4 hours (treatment period 2). There will be a 1-2 hour preparatory washout phase prior to treatment period 1 and another 1-2 hour washout between treatment period 1 and 2. Infants will be monitored for a further 12-hours post-completion of the crossover trial for safety events.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-Short PRT Sequence (Experimental): Long PRT set during first treatment period; Short PRT set during second treatment period
  Interventions: Other: Long PRT; Other: Short PRT
- Short-Long PRT Sequence (Experimental): Short PRT set during first treatment period; Long PRT set during second treatment period
  Interventions: Other: Long PRT; Other: Short PRT

INTERVENTIONS:
Other: Long PRT — PRT (in seconds) set at 75% of inspiratory time (in seconds)
  Other Names: Long Pressure Rise Time
Other: Short PRT — PRT (in seconds) set at 33% of inspiratory time (in seconds).
  Other Names: Short Pressure Rise Time

SUMMARY:
Babies born extremely preterm (<28 weeks of pregnancy) require support to breathe. Some babies require help to breathe from a breathing machine (mechanical ventilator). While this keeps babies alive, it may damage their lungs. To reduce this damage, doctors and nurses take particular care to try and provide the gentlest breathing support possible. However, evidence is still required to determine how to best support babies' breathing, whilst preventing lung damage and longer-term lung problems.

This clinical trial aims to compare two ways of adjusting a common setting on the breathing machine. This setting is called the pressure rise time or PRT. The PRT determines how quickly the breathing machine inflates a premature baby's lungs. A short PRT quickly inflates the lungs. A long PRT inflates the lungs more slowly. Previous research suggests that more slowly inflating the baby's lungs may cause less lung damage and still allow oxygen to be delivered to and carbon dioxide to be cleared from the lungs. However, larger studies are required to determine whether this should become the standard treatment.

This study investigates whether inflating the baby's lungs more slowly (long PRT) using the breathing machine is as effective as the PRT setting currently used (short PRT, more quickly inflating the lungs).

The main question it aims to answer is: Does how quickly the breathing machine inflates an extremely preterm baby's lung impact their oxygen levels?

DETAILED DESCRIPTION:
The FLOW-VENT trial will investigate if using a long pressure rise time (PRT; thereby reducing the speed of gas flow) compared to a short PRT, during synchronised, patient-triggered, volume-targeted conventional mechanical ventilation in extremely preterm infants within the first postnatal week impacts an infant's oxygenation.

All infants born extremely preterm (<28 weeks' gestation) require breathing support to survive. However, this support can damage their lungs. Rates of bronchopulmonary dysplasia (BPD), the chronic lung disease of extreme prematurity, are increasing. This is despite 'lung protective' respiratory support and ventilation strategies that aim to minimise harm to the preterm lung.

Pre-clinical evidence suggests that gas flows lower than currently used during respiratory support of these infants may be a major, and easily modifiable way of reducing preterm lung injury (Tingay 2024; Bach 2012). Current guidelines lack evidence for suggested gas flow settings. Many ventilators now modulate ventilator gas flows by a setting known as pressure rise time (PRT).

FLOW-VENT is a prospective, multicentre, unblinded, randomised crossover trial enrolling 68 extremely preterm infants born <28 weeks gestational age. A long PRT is defined as a PRT set at 75% of the inspiratory time (Ti). A short PRT is defined as a PRT set at 33% of the Ti.

Given the crossover design, infants will receive both the long and short PRT setting. Extremely preterm infants will be randomised to a 'sequence' which will determine the order in which they are exposed to the different PRTs; either:

* Long-Short PRT Sequence: Long PRT in the first treatment period and Short PRT in the second treatment period, OR
* Short-Long PRT Sequence: Short PRT in the first treatment period and Long PRT in the second treatment period.

The trial crossover phase (~10-12 hours) consists of: 1) Preparatory washout period (1 to 2 hours); 2) First treatment period (4-hours); 3) Washout period (1 to 2 hours); 4) Second treatment period (4-hours). Following this, there is a 12-hour follow-up period to monitor for adverse/safety events. The primary outcome (average S/F ratio) is assessed only during the 4-hour treatment periods.

Results from this trial will inform the decision to proceed to a larger randomised trial, powered for longer term respiratory outcomes (e.g. time to extubation from mechanical ventilation, BPD at 36 weeks' postmenstrual age).

ELIGIBILITY:
Inclusion Criteria:

* Admitted to participating neonatal intensive care unit
* Born between 22+0 to 27+6 weeks' gestation
* Current weight ≥400 grams
* Receiving synchronised, patient-triggered, volume-targeted (all breaths) conventional mechanical ventilation (Pressure Control-Assist Control + Volume Guarantee [PC-AC+VG] mode on Dräger Babylog VN500/800 ventilators) initiated within 72-hours post birth
* Postnatal age ≥6 hours and ≤7 days
* Received surfactant therapy
* Clinically stable (as per treating and research team consensus)
* Parent(s)/legal guardian provides prospective informed consent.

Exclusion Criteria:

* Major congenital anomaly involving the cardiac, respiratory or gastrointestinal systems, or a known genetic syndrome or diagnosis that might affect respiratory course and outcomes
* Severe pulmonary hypoplasia due to anhydramnios or oligohydramnios before 22 weeks in which the neonatal consultant anticipates that pulmonary hypoplasia related respiratory failure will be the major respiratory problem in early postnatal life
* Receiving (or expected to receive within the next 12 hours) any other mode of mechanical ventilation including synchronised intermittent mandatory ventilation (SIMV), pressure support ventilation (PSV) or high-frequency oscillatory ventilation
* Planned for extubation from mechanical ventilation within the next 12 hours.

Ages: 6 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in peripheral oxygen saturation to fraction of inspired oxygen ratio (S/F Ratio) measured each minute during each treatment period (0 minutes to 4 hours) | 0 minutes then each minute up to 4 hours for each of the Long PRT and Short PRT 4-hour treatment periods

SECONDARY OUTCOMES:
Change in pressure rise time (PRT) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in mean airway pressure (MAP) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during of the Long PRT and Short PRT 4-hour treatment periods.
Change in positive end expiratory pressure (PEEP) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in peak inspiratory pressure (PIP) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in tidal volume (VT) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in respiratory rate measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in minute ventilation measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in endotracheal tube leak measured each minute during each treatment period (0 minutes to 4 hours) | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in inspiratory time (Ti) measured each minute during each treatment period (0 minutes to 4 hours) | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in inspiratory gas flows measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in peripheral oxygen saturation (SpO2) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in fraction of inspired oxygen (FiO2) measured each minute during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Change in incidence of significant oxygen desaturation measured during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
  Significant oxygen desaturation is defined as SpO2 <80% for >30 seconds
Change in total number FiO2 changes measured during each treatment period (0 minutes to 4 hours). | Measured during each of the Long PRT and Short PRT 4-hour treatment periods.
Incidence of air leak (pneumothorax or pneumomediastinum) | Completed for each participant at end of their study period: 22-24 hours from study commencement.
Incidence of pulmonary haemorrhage receiving management (increased PEEP/PIP/FiO2 or blood products) | Completed for each participant at end of their study period: 22-24 hours from study commencement.
Incidence of resuscitation (defined as receiving external cardiac compressions or adrenaline boluses) | Completed for each participant at end of their study period: 22-24 hours from study commencement.
Incidence of death | Completed for each participant at end of their study period: 22-24 hours from study commencement.
Incidence of treating consultant request to discontinue randomly allocated PRT prematurely | Completed for each participant at end of their study period: 22-24 hours from study commencement.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin N Ferguson, BSc MBBS, Principal Investigator — Murdoch Childrens Research Institute
Locations (3):
- Australia (3):
  - Mercy Hospital for Women, Heidelberg, Victoria
  - The Royal Women's Hospital, Parkville, Victoria
  - Joan Kirner Women's and Children's Hospital, Saint Albans, Victoria

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data set collected for this analysis of the FLOW-VENT trial will be available six months after publication of the primary outcome, if the below access criteria are met.
  The study protocol, statistical analysis plan and consent forms will also be available. The data may be obtained from the Murdoch Children's Research Institute (MCRI) by emailing kristin.ferguson@mcri.edu.au, david.tingay@rch.org.au and mctc@mcri.edu.au.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after publication of primary outcome.
Access Criteria: Prior to releasing any data the following are required:
  1. A Data Transfer Agreement must be signed between relevant parties.
  2. The MCRI Sponsorship Committee must review and approve your protocol and statistical analysis plan which must include and describe how the data will be used and analysed.
  3. An Authorship Agreement to be agreed to and signed between relevant parties. The Agreement must include details regarding appropriate recognition. Authorship may not be justifiable but some form of acknowledgement is requested.
  4. Agreement to cover any additional costs relating to the provision of the data.
  5. Evidence of ethics approval or waiver of approval, to be compliant with the data transfer agreement and ethics requirements at our end.
  Data will only be shared with a recognised research institution where the MCRI Sponsorship Committee has approved the proposed analysis plan.
URL: https://www.mcri.edu.au/research/core-facilities-services/melbourne-children-trials-centre

REFERENCES:
- [Background] Tingay DG, Fatmous M, Kenna K, Chapman J, Douglas E, Sett A, Poh QH, Dahm SI, Quach TK, Sourial M, Fang H, Greening DW, Pereira-Fantini PM. Speed of lung inflation at birth influences the initiation of lung injury in preterm lambs. JCI Insight. 2024 Aug 6;9(18):e181228. doi: 10.1172/jci.insight.181228. PMID 39106107
- [Background] Sherer JL. Survey highlights the occupational hazards of nursing. Hospitals. 1993 May 20;67(10):60. No abstract available. PMID 8491472
- [Background] Bach KP, Kuschel CA, Oliver MH, Bloomfield FH. Ventilator gas flow rates affect inspiratory time and ventilator efficiency index in term lambs. Neonatology. 2009;96(4):259-64. doi: 10.1159/000220765. Epub 2009 May 27. PMID 19478530
- [Background] Riley M. Testimony of the American Society for Microbiology before the House Subcommittee on Investigations and Oversight, House Subcommittee on Natural Resources, Agriculture Research and Environment, and the House Subcommittee on Science, Research and Technology of the House Committee on Science and Technology. Hearing on "The coordinated framework for the regulation of biotechnology", July 23, 1986. Recomb DNA Tech Bull. 1986 Sep;9(3):151-61. No abstract available. PMID 3466239
- [Background] Chong D, Kayser S, Szakmar E, Morley CJ, Belteki G. Effect of pressure rise time on ventilator parameters and gas exchange during neonatal ventilation. Pediatr Pulmonol. 2020 May;55(5):1131-1138. doi: 10.1002/ppul.24724. Epub 2020 Mar 9. PMID 32150670